CLINICAL TRIAL: NCT05269433
Title: The Effect of Attention Training on Symptoms and Emotion Regulation in Depressive Patients: Validation of the Online Contingent Attention Training (OCAT).
Brief Title: The Effect of Attention Training on Symptoms and Emotion Regulation in Depressive Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Alexianen Zorggroep Tienen (Unknown); Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0G054-2021-07
Record Dates: First submitted 2022-02-11; First posted 2022-03-08 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Depression
Keywords: Emotion Regulation; Attention Training; Psycho-education; Depression
MeSH Terms: conditions — Depression; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PSE + OCAT-sham (Active Comparator): Psycho-education video + an active placebo training consisting of 10 sessions of ±12 minutes each (during an intervention period of two weeks) will be administered. The training task is an undirected scrambled sentences task with online contingent feedback (only) on the speed with which the sentences were made. In this condition, participants will not receive feedback on emotional attention.
  Interventions: Behavioral: OCAT-sham; Other: Psycho-education video
- PSE + OCAT (Experimental): Psycho-education video + an attention training consisting of 10 sessions of ±12 minutes each (during an intervention period of two weeks) will be administered. The training task is a positively directed scrambled sentences task with online contingent feedback on how much attention was paid to positive vs. negative words (emotional attention), along with feedback on the speed with which the sentences were made.
  Interventions: Behavioral: OCAT; Other: Psycho-education video
- PSE + OCAT+ (Experimental): Psycho-education video + short motivational video before each training session + an attention training consisting of 10 sessions of ±12 minutes each (during an intervention period of two weeks) will be administered. The training task is a positively directed scrambled sentences task with online contingent feedback on how much attention was paid to positive vs. negative words (emotional attention), along with feedback on the speed with which the sentences were made.
  Interventions: Behavioral: OCAT; Other: Psycho-education video; Other: Motivational video

INTERVENTIONS:
Behavioral: OCAT-sham — Placebo version of the online contingent attention training preceded by a psycho-education movieclip.
  Arms: PSE + OCAT-sham
Behavioral: OCAT — Online contingent attention training preceded by a psycho-education movieclip.
  Arms: PSE + OCAT; PSE + OCAT+
Other: Psycho-education video — All groups watch a psycho-education video before the start of the 10-day attention training.
Other: Motivational video — Participants in the OCAT+ condition watch a short motivational video before each training session.
  Arms: PSE + OCAT+

SUMMARY:
Attention control for external information and cognitive control for internal information play a causal role in emotion regulation according to different theories and research. Prior research shows that an interactive attention control training in which participants learn to unravel scrambled sentences ("life is my a party mess") in a positive manner ("my life is a party") by receiving feedback on their eye movements while attending to the valenced words, can facilitate participants to be more able to re-interpret negative information in a positive manner. In the current study we want to test the effect of psycho-education in combination with a 10 day attention control training to see if this has a positive effect on depressive, anxiety and stress symptoms, emotion regulation and self-esteem in depressed patients. The study takes place in a psychiatric hospital (Alexianen Zorggroep Tienen) while participants are staying there to receive treatment.

DETAILED DESCRIPTION:
Attention control for external information and cognitive control for internal information play a causal role in emotion regulation according to different theories and empirical research. Former research in the lab of the investigators has shown positive effects of an interactive attention control training where participants learned to unscramble scrambled sentences ("life is my a party mess") in a positive way ("my life is a party") by getting eye-tracking feedback about attention for positive ("party") vs. negative information ("mess") when looking at the sentences. After the training, participants could better reinterpret negative pictures in a positive way. Attention- and cognitive control mechanisms prior to negative stressors (proactive control) and after negative stressors (reactive control) may play a role in the effects. Research suggests that low perceived control and negative expectations about future emotion regulation skills results in lower proactive control and a higher need of reactive control. Based on this, the assumption can be made that the effects of attention control training - targeting reactive control - could benefit from adding techniques that affect proactive control (i.e. psycho-education, additional short motivational video). In the present study this is investigated by testing a new 10 day attention control training to see if this has a positive effect on depressive, anxiety and stress symptoms, emotion regulation and self-esteem. Participants between 18 to 65 years of age are recruited during their admission in a psychiatric hospital (Alexianen Zorggroep Tienen). The attention control training is a new smartphone based application where participants are asked to unscramble scrambled sentences into grammatically correct sentences. Participants are randomly assigned to one of three conditions: a training condition with preceding psycho-education video (OCAT), a control condition with preceding psycho-education video (OCAT-sham), and a training condition with preceding psycho-education video and additional short motivational video before each training session (OCAT+). In the training conditions (OCAT and OCAT+), participants are asked to unscramble the scrambled sentences in a positive way. By swiping, participants can see parts of the sentences. This gives the investigators an image about the processing of the sentences. This procedure allows to measure how long participants attend to positive and negative words. In the training conditions participants receive feedback about the duration of processing positive and negative words. In the control group participants unscramble the sentences as fast as possible without feedback on emotional attention. Participants in the control condition only receive feedback about the speed by which the sentences are unscrambled. Before and after the 10 training sessions, attention of the participants is measured. Questionnaires on depressive, anxiety, and stress symptoms, emotion regulation strategies, and self-esteem are administered before and after the training. Moreover, participants' credibility and expectancy towards the training will also be measured. There is also a follow-up measure 3 months after the training. All groups (training and control) watch a psycho-education video before the start of the training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depressive disorder
* Admission to a psychiatric hospital (Alexianen PK, Tienen)

Exclusion Criteria:

* Current psychotic disorder
* Current neurological impairments
* Current alcohol addiction
* Current treatment with antidepressants that has not yet been kept constant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in depression symptoms | pre-test (before starting the training), post-test (immediately after the training), follow-up (three months after the training)
  Measured by the Depression and Anxiety Stress Scale (DASS-21), a self report questionnaire containing 21 items to measure the severity of a range of common symptoms for depression, anxiety and stress. Participants are required to indicate the presence of a symptom over the previous week. Each item of the questionnaire is scored from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Higher scores indicate more symptoms. The questionnaire comprises three subscales (Depression, Anxiety, and Stress). For this specific outcome measure, the depression subscale will be used (7 items) to investigate the specific effects of the training on depressive symptoms.
Changes in anxiety symptoms | pre-test (before starting the training), post-test (immediately after the training), follow-up (three months after the training)
  Measured by the Depression and Anxiety Stress Scale (DASS-21), a self report questionnaire containing 21 items to measure the severity of a range of common symptoms for depression, anxiety and stress. Participants are required to indicate the presence of a symptom over the previous week. Each item of the questionnaire is scored from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Higher scores indicate more symptoms. The questionnaire comprises three subscales (Depression, Anxiety, and Stress). For this specific outcome measure, the anxiety subscale will be used (7 items) to investigate the specific effects of the training on anxiety symptoms.
Changes in stress symptoms | pre-test (before starting the training), post-test (immediately after the training), follow-up (three months after the training)
  Measured by the Depression and Anxiety Stress Scale (DASS-21), a self report questionnaire containing 21 items to measure the severity of a range of common symptoms for depression, anxiety and stress. Participants are required to indicate the presence of a symptom over the previous week. Each item of the questionnaire is scored from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Higher scores indicate more symptoms. The questionnaire comprises three subscales (Depression, Anxiety, and Stress). For this specific outcome measure, the stress subscale will be used (7 items) to investigate the specific effects of the training on stress symptoms.

SECONDARY OUTCOMES:
Changes in cognitive emotion regulation strategies | pre-test (before starting the training), post-test (immediately after the training), follow-up (three months after the training)
  Measured by the Cognitive Emotion Regulation Questionnaire (CERQ), a self-report questionnaire measuring different emotion regulation strategies, containing 36 items with a 5-point Likert response format scored from 1 ("Almost never") to 5 ("Almost always"). This questionnaire has 9 sub-scales: self-blame, other-blame, rumination, catastrophizing, putting into perspective, positive refocusing, positive reappraisal, acceptance and refocus on planning. Each sub-scale has a scoring range between 4 and 20. A higher score represents a greater frequency of engaging in that emotion regulation strategy.
Self-Esteem | pre-test (before starting the training), post-test (immediately after the training), follow-up (three months after the training)
  Measured by the Rosenberg Self Esteem Scale (RSES), a self-report questionnaire assessing global self-esteem. The questionnaire consists of 10 items with five positively worded items and five negatively worded. Four response categories are used, with items scored from 0 (Strongly Disagree) to 3 (Strongly Agree).
Treatment Credibility and Expectancy | pre-test (before starting the training), post-test (immediately after the training)
  Measured by the Credibility/Expectancy Questionnaire (CEQ). It measures participants' credibility and expectancy of the training. In the credibility scale, 4 items are rated on 9-point scales ranging from 1 (Not at all logical/useful/confident) to 9 (Very logical/effective/confident). This leads to a total score on this scale between 3 and 27. In the expectancy scale (2 items) the same 9-point scale is used, along with an 10-point scale (from 1% to 100%). Responses are standardized to get the total expectancy score. Higher scores represent higher credibility and expectancy. In this version of the CEQ, an extra item is included containing the question if the participant believes to be part of the placebo condition (to be responded with 'yes/no').
Changes in emotional attention | pre-test (before starting the training), post-test (immediately after the training)
  Measured by a baseline measure in the OCAT app. Participants perform a Scrambled Sentences Task to measure pre-post changes in emotional attention biases. Participants are instructed to unscramble the sentences as fast as possible to form the first grammatically correct and meaningful positive or negative sentence that spontaneously came to their mind, using only 5 words.
  Participants are asked to press a fixation cross to start the reading section of the SST. Then, 6 words are hidden into individual squares and participants move their fingers to uncover and read the corresponding word. When participants move their fingers away from one word to the position of another word, the previous word is hidden again and the next word is shown. The position and coordinates of the participants' finger on the screen allow us to monitor the exact time that participants are attending and reading each word, and thus to measure attention biases towards negative and positive words.

CONTACTS AND LOCATIONS:
Overall Officials: Rudi De Raedt, Professor, Principal Investigator — University Ghent
Locations (3):
- Belgium (3):
  - Ghent University, Ghent, Oost-Vlaanderen
  - Alexianen PK Zorggroep Tienen, Tienen, Vlaams-Brabant
  - KARUS, Sint-Denijs-Westrem

IPD SHARING:
Plan to Share IPD: No
* Individual participant data will not be available.
  * Other documents will be available: Statistical Analysis Plan, Study Protocol (upon request to the researchers).

REFERENCES:
- [Background] Sanchez-Lopez A, Everaert J, Van Put J, De Raedt R, Koster EHW. Eye-gaze contingent attention training (ECAT): Examining the causal role of attention regulation in reappraisal and rumination. Biol Psychol. 2019 Mar;142:116-125. doi: 10.1016/j.biopsycho.2019.01.017. Epub 2019 Feb 5. PMID 30735680
- [Background] De Raedt R, Hooley JM. The role of expectancy and proactive control in stress regulation: A neurocognitive framework for regulation expectation. Clin Psychol Rev. 2016 Apr;45:45-55. doi: 10.1016/j.cpr.2016.03.005. Epub 2016 Mar 24. PMID 27064551